CLINICAL TRIAL: NCT02598323
Title: Premature Labour Screening by Cervical Ultrasound for Asymptomatic Pregnant Women in the PACA Region. Various Treatment Strategies : 1. Progesterone 200mg (Vaginal Way) 2. Pessary 3. Vaginal Stitching 4. Rest
Brief Title: Prevention and Treatment of Premature Labour for Asymptomatic Pregnant Women
Acronym: Echo-col
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2014-24; AP-HM (Registry Identifier: RCAPHM14_0191)
Record Dates: First submitted 2015-11-04; First posted 2015-11-05 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-11

CONDITIONS: Premature Labour
MeSH Terms: conditions — Obstetric Labor, Premature | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- patients with active singleton pregnancy between 16 and 26 SA (Experimental)
  Interventions: Device: ultrasound

INTERVENTIONS:
Device: ultrasound

SUMMARY:
State of the question and research objective: International trials have shown that ultrasound measurement of the cervix identifies a population at high risk of preterm delivery. In case of short neck several types of treatments can be recommended: progesterone, the establishment of a strapping or pessary. These three treatments reduce the risk of preterm delivery. There is no French study.

The objective of this study is to reduce prematurity in the PACA region Monaco-Corsica by introducing a routine ultrasound screening strategy asymptomatic short necks.

Population concerned: All patients with active singleton pregnancy between 16 and 26 SA SA are eligible to ultrasound of the cervix.

* Primary endpoint: delivery rate before 37 weeks.
* Criteria secondary judgments rate of deliveries before 37 weeks, neonatal mortality morbidity.

Expected result: a prematurity of 50%

DETAILED DESCRIPTION:
State of the question and research objective: International trials have shown that ultrasound measurement of the cervix identifies a population at high risk of preterm delivery. In case of short neck several types of treatments can be recommended: progesterone, the establishment of a strapping or pessary. These three treatments reduce the risk of preterm delivery. There is no French study.

The objective of this study is to reduce prematurity in the PACA region Monaco-Corsica by introducing a routine ultrasound screening strategy asymptomatic short necks.

Expected result: a prematurity of 50%

Population concerned: All patients with active singleton pregnancy between 16 and 26 SA SA are eligible to ultrasound of the cervix.

Method of observation and deduction investigation: Study before / after comparing two periods: period A (2013) and Period B (2015).

* Primary endpoint: delivery rate before 37 weeks.
* Criteria secondary judgments rate of deliveries before 37 weeks, neonatal mortality morbidity.

Data flow mode:

Duration and terms of organization of research: The actual duration of the study (preparation and implementation, monitoring and inclusions) is set at 36 months. This study will be conducted in the context of networks. All maternity hospitals belonging to these networks will be invited to participate. Referents investigating doctors will be appointed.

The attaché of clinical research in collaboration with the Network Coordinator, Michele Marcot, get back the data for the year 2013 by the transfer records examination, delivery specifications, reviews of the hospitalization mother and child.

Data collection for 2015 will be based on a collection form that will complement the investigators involved in the project at the inclusion of the patient.

These sheets will be collected in real time by the RCAF in charge of monitoring the study will proceed to their seizure.

Positive cases (short necks - less than 25mm) will be offered or not progesterone treatment, banding or the establishment of a pessary according to the habits of the practitioner and the service protocol.

If treatment with progesterone is retained, it is Vaginal Progesterone 200mg, natural micronized progesterone without excipients with known effect in capsule form.

Data Analysis Method: Statistical analysis will be initiated only after verification of the validity of the database (queries broadcast from clinicians involved in the study, consistency checks). There is a procedure and data anonymization algorithm giving each individual a number. A lookup table is available, separate from the operating base. Only the number will be entered into the computer database. The database will then be frozen. After the base gel, the consolidated data will be processed by the statistician. Data analysis will be performed using the SPSS Version 17.0 software for Windows by the statistician of the Unit for Clinical Research Methodology (Loundou Anderson, head Prof. Pascal Auquier).

Statistical significance tests will be set at 5%. The type of unilateral or bilateral test will depend on the chosen alternative, especially based on the results already available in previous studies.

The qualitative variables are expressed in terms of numbers and percentages, and quantitative variables will be reported using the usual parameters of position (mean, median) and dispersion (standard deviation, range). The normality of the distributions of quantitative data will be systematically searched using the Shapiro-Wilks test. If variables are not normally distributed, conventional processing techniques (logarithmic, ...) will be implemented.

Initially, a comparability study populations for inclusion will be made on all the variables collected at that time: socio-demographic and clinical (using Mantel-Haenszel test, the Chi-2 or accurate Fisher for qualitative variables, and Student's t test or ANOVA for quantitative variables) to reveal potential confounding factors to consider when analyzing the criteria of judgment. Comparisons between the study populations will also be conducted on all the criteria of secondary judgments. Adjustments will be made on the variables identified as confounding factors by conducting multivariate analysis (analysis of variance, multivariate logistic regression).

Justification of the number of subjects or power analysis: The prematurity rate was 7.4% in 2013 in France (PACA, Périnat data 2010).

We expect a reduction in this rate of 1.5 points (or 6%) over the period 2015 referring to the reduction of prematurity obtained by Kiss, et al, 2003.

To achieve this reduction in preterm birth rate, include 3500 patients in each period. Considering the selection criteria and the active files of the various partners, the inclusion of patients in the period 3500 2014 is quite achievable.

(44,000 births per year at the network level, among which are ensuring that 10% of them meet the predefined criteria). Regarding the second period, the reasoning is the same; among the list of eligible patients, a random draw will be conducted to determine the 3500 patients representing this period. Thus for 3500 patients included in the period 2014, 10% will have a short neck or 350 patients who will be offered the Progesterone, a banding or the establishment of a pessary.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years,
* pregnancy with single fetus,
* gestational age between 16SA and 26SA,
* asymptomatic patients, that is to say, without sign of preterm labor layout

Exclusion Criteria:

* Maternal Pathology (Pre Eclampsia, non-insulin dependent diabetes, insulin dependent gestational diabetes or unbalanced)
* uterine malformation
* fetal malformation or fetal chromosomal abnormality
* premature Work in Progress (cervix dilated to more than 2 cm or regular uterine contractions and felt)
* Signs of chorioamnionitis
* Allergy to progesterone
* Taking progesterone in the month preceding the inclusion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3500 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
delivery rate before 37 weeks | 21 weeks maximum

SECONDARY OUTCOMES:
neonatal mortality | about 30 weeks
rate of newborns admitted to intensive care in the first month of life | about 30 weeks
length of stay in intensive care | about 30 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Urielle Desalbres, Study Director — AP-HM
Locations (1):
- AP-HM, Marseille, France

REFERENCES:
- [Derived] Figarella A, Chau C, Loundou A, d'Ercole C, Bretelle F. The introduction of a universal transvaginal cervical length screening program is associated with a reduced preterm birth rate. Am J Obstet Gynecol. 2023 Feb;228(2):219.e1-219.e14. doi: 10.1016/j.ajog.2022.07.046. Epub 2022 Aug 4. PMID 35932876